CLINICAL TRIAL: NCT04370795
Title: Matched Related and Unrelated Donor Stem Cell Transplantation for Severe Combined Immune Deficiency (SCID): Busulfan-based Conditioning With h-ATG, Radiation, and Sirolimus
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200037; 20-I-0037
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Severe Combined Immune Deficiency (SCID)
Keywords: Post-Transplant; Hematopoietic; Allogeneic; Graft-Versus-Host Disease; Irradiation
MeSH Terms: conditions — Severe Combined Immunodeficiency; Graft vs Host Disease | interventions — Sirolimus; Busulfan; Granulocyte Colony-Stimulating Factor; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients will be treated with Total Body Irradiation (TBI)
  Interventions: Drug: Sirolimus; Drug: Busulfan; Drug: Horse -Anti-thymocyte; Drug: G-CSF; Radiation: Total Body Irradiation (TBI)
- Group 2 (Active Comparator): Patients will not be treated with Total Body Irradiation (TBI)
  Interventions: Drug: Sirolimus; Drug: Busulfan; Drug: Horse -Anti-thymocyte; Drug: G-CSF

INTERVENTIONS:
Drug: Sirolimus — Post transplant immunosuppressant drug
Drug: Busulfan — Conditioning drug
Drug: Horse -Anti-thymocyte — Immune suppression conditioning drug
Drug: G-CSF — Used to prevent infection and neutropenic fevers caused by chemotherapy
Radiation: Total Body Irradiation (TBI) — Conditioning (only patients in Group 1 will receive TBI)
  Arms: Group 1

SUMMARY:
Background:

Severe combined immune deficiency (SCID) is a group of conditions where the immune system does not work properly. The only cure for most SCIDs is a stem cell transplant (getting cells from a donor). These transplants can have serious complications. Before the transplant, people often get high doses of drugs and radiation to prepare the body to accept the cells from the donor. Researchers want to see if low doses of drugs alone without radiation work just as well as low doses of drugs with radiation for SCID patients getting stem cell transplants.

Objective:

To test a set of drugs with or without radiation given before a stem cell transplant.

Eligibility:

People ages 3-40 who have SCID and who have a stem cell donor - either related or unrelated.

Design:

Participants will be admitted to the hospital 10 days before transplant. They will undergo:

medical history

medication review

physical exam

blood and urine tests (may include a 24-hour urine collection)

heart, lung, and breathing tests

imaging scans

bone marrow sample

nutrition assessment

dental exam

eye exam

meeting with a social worker.

Participants will get a plastic port called a central line. It is a hollow tube that is placed in the upper chest. It will be used to give medicines and take blood.

All participants will take chemotherapy drugs. Some will get radiation.

Participants will have a stem cell transplant. They will get the cells as an infusion through their central line. They will stay in the hospital for 30 days after transplant.

Participants must stay within 1 hour of NIH for 3 months after transplant. During this time, they will have follow-up visits at NIH at least once a week. Then they will have follow-up visits once or twice a year for 5-6 years.

DETAILED DESCRIPTION:
This is an open-label pilot study of human leukocyte antigen (HLA)-matched related and unrelated donor hematopoietic stem cell (HSC) transplant (also referred to as peripheral blood stem cell [PBSC] transplant or bone marrow transplant [BMT]) for up to 20 patients with severe combined immune deficiency (SCID). SCID is most commonly caused by mutations in the IL2RG gene encoding the interleukin (IL) receptor signaling gamma chain (gamma c); however, patients with JAK-3 mutations have the same phenotypes and are similarly affected. The study population is older children (greater than or equal to 3 years of age) and adults (less than or equal to 40 years of age) who are experiencing deteriorating and/or dysfunctional immunity and/or any of a constellation of severe or chronic medical problems warranting transplantation. The study is designed to evaluate whether the use of uniquely designed transplant conditioning either containing total body irradiation (TBI) or not, along with a graft-versus-host disease (GvHD) prevention regimen achieves sufficient engraftment of donor HSCs to facilitate robust restoration of cellular immunity (T cell/natural killer [NK] cell number and function) including thymic function, and humoral immunity (B cell number and function), while at the same time enhancing tolerance of the donor graft in a fashion that reduces the occurrence of GvHD but not significantly enhancing the risk of post-transplant viral infection. One target population is SCID patients who received matched sibling or haploidentical lymphocyte-depleted transplants as infants with little or no myeloid conditioning, resulting in variable restoration of T cell immunity, but little or no restoration of NK or B cell immunity. Another target population is SCID patients with partial production or function of gamma c or JAK3 or SCID patients with clonal somatic reversion of the mutation in the IL2RG or JAK-3 gene, who have less severe immune deficiency in childhood. A subset of patients from all of these target SCID populations may experience progressive deterioration of immune function leading to acute and chronic medical problems that warrant consideration of allogeneic transplant to restore immunity.

The conditioning and GvHD prevention regimens for this HSC transplant protocol are designed to use mobilized PBSCs or bone marrow (if mobilization is not possible) from either an HLA-matched related donor (MRD) as first choice or from an HLA-matched unrelated donor (MUD) for those without an appropriate HLA-MRD. If there is no appropriate MRD nor MUD adult donor available, then an appropriate cord blood from the cord blood registries may be used for small children SCID recipients. We propose using a busulfan-based, nonmyeloablative conditioning regimen plus or minus TBI combined with horse anti-thymocyte globulin (h-ATG) immune suppression conditioning plus post-transplant sirolimus as a tolerance-inducing immunosuppressant to prevent GvHD.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have confirmed genetic diagnosis of SCID (gamma c or JAK3 deficiency) by identification of a mutation in the responsible genes or by demonstrating failure to detect gamma c or JAK3 in immune blood cells (as in the case of patients who have been treated but now have waning immunity).
* Must have either evidence of waning immunity by T cell analysis, and/or sufficient complications from underlying disease to warrant undergoing transplantation as defined as meeting greater than or equal to1 of the following clinical criteria:

  i- Infections (not including molluscum, warts, or mucocutaneous candidiasis; see vii and viii below): 3 significant new or chronic active infections during the 2 years preceding evaluation for enrollment, with each infection accounting for one criterion.

Infections are defined as an objective sign of infection (fever >38.3 (Infinite)C [101 degrees F] or neutrophilia or pain/redness/swelling or radiologic/ultrasound imaging evidence or typical lesion or histology or new severe diarrhea or cough with sputum production). In addition to one or more of these signs/symptoms of possible infection, there also must be at least 1 of the following criteria as evidence of the attending physician s intent to treat a significant infection (a and b) or objective evidence for a specific pathogen causing the infection (c):

1. Treatment (not prophylaxis) with systemic antibacterial, antifungal or antiviral antibiotics for greater than or equal to 14 days; OR
2. Hospitalization of any duration for infection; OR
3. Isolation of a bacteria, fungus, or virus from biopsy, skin lesion, blood, nasal washing, bronchoscopy, cerebrospinal fluid or stool likely to be an etiologic agent of infection.

ii. Chronic pulmonary disease as defined by:

1. Bronchiectasis by x-ray computerized tomography; OR
2. Pulmonary function test (PFT) evidence for restrictive or obstructive disease that is less than or equal to 60% of predicted for age; OR
3. Pulse oximetry less than or equal to 94% in room air (if patient is too young to comply with performance of PFTs).

iii. Gastrointestinal enteropathy:

1. Diarrhea-watery stools greater than or equal to 3 times per day (of at least 3 months duration that is not a result of infection as defined in criterion # i. above); OR
2. Endoscopic evidence (gross and histologic) for enteropathy (endoscopy will only be performed if medically indicated); OR
3. Other evidence of enteropathy or bacterial overgrowth syndrome, including at least one of the following: malabsorption of fat soluble vitamin(s), abnormal D-xylose absorption, abnormal hydrogen breath test, or evidence of protein-losing enteropathy (for example, increasingly high or frequent dosing of IV gamma globulin supplement required to maintain blood IgG level).

iv. Poor nutrition: Requires G-tube or IV feeding supplement to maintain weight or nutrition.

v. Auto- or allo-immunity: Objective physical findings including but are not limited to at least one of the following: alopecia, severe rashes, uveitis, joint pain with redness or swelling or limitation of movement that is not a result of infection, lupus-like lesions, and granulomas (not including auto- or alloimmune enteropathy, which is criterion iii). Where possible and appropriate, diagnosis will be supported by histopathology or another diagnostic modality.

vi. Failure to grow in height: less than or equal to 3rd percentile for age.

vii. Skin molluscum contagiosum OR warts (this criterion is satisfied if molluscum consists of greater than or equal to 10 lesions or there are greater than or equal to 2 lesions at each of two or more widely separated anatomic sites; or there are greater than or equal to 3 warts at different anatomic sites at the same time; or the patient has both molluscum and warts).

viii. Mucocutaneous candidiasis (chronic oral thrush or candida esophagitis or candida intertriginous infection or candida nail infection; must be culture positive to satisfy this criterion).

ix. Hypogammaglobulinemia: Requires regular IgG supplementation.

* Aged 3-40 years, inclusive.
* Must have a 6/6 HLA-MRD graft available, or an HLA-matched unrelated PBSC graft (10/10 or 9/10 mismatch) available, or a minimum of 4/6 HLA-matched cord blood product available (if the cord blood graft is less than 5.0x10(7) cells, a second appropriate 4/6 or greater match cord blood product must be available).
* Mismatched MUD and Cord Blood transplants need to have Class I and II HLA antibody screen, DSA should be avoided.
* Must be HIV negative.
* Must be able to stay within 1 hour s travel of the NIH for the first 3 months after transplantation and have a family member or other designated companion to stay with during the post-transplant period.
* Must provide a durable power of attorney (DPA) for health care decisions to an appropriate adult relative or guardian in accordance to NIH-200 NIH Advance Directive for Health Care and Medical Research Participation .
* For participants of reproductive potential, must agree to consistently use highly effective contraception throughout study participation and for at least 3 months after the study.

Acceptable forms of contraception are:

a. For females:

i. Condoms, male or female, with or without a spermicide;

ii. Diaphragm or cervical cap with spermicide;

iii. Intrauterine device;

iv. Contraceptive pills or patch, Norplant, Depo-Provera, or other FDA-approved contraceptive method;

v. Male has previously undergone a vasectomy.

b. For males: Condoms or other contraception with partner.

EXCLUSION CRITERIA:

1. Eastern Cooperative Oncology Group (ECOG) or equivalent performance status of 3 or more (see ECOG performance status guidelines, available at https://ecog-acrin.

   org/resources/ecog-performance-status).
2. Left ventricular ejection fraction <40%.
3. Transaminases >5x upper limit of normal based on the patient s clinical situation and at the discretion of the investigator.
4. Liver alkaline phosphatase >10x upper limit of normal based on the patient s clinical situation and at the discretion of the investigator.
5. Psychiatric disorder or mental deficiency severe enough as to make compliance with the BMT treatment unlikely, and/or making informed consent impossible.
6. Major anticipated illness or organ failure incompatible with survival from alloPBSC, MUD, or unrelated cord blood transplant.
7. Uncontrolled seizure disorder.
8. Any condition that, in the opinion of the investigator, contraindicates participation in this study.
9. Pregnant or lactating females.

INCLUSION OF VULNERABLE PARTICIPANTS

Children: Children 3 years of age and older may enroll on this study because the condition under study affects children and the study holds the prospect for direct benefit.

Pregnant and Lactating Women: Pregnant women are excluded from this study due to risks associated with the study intervention and the effects of the combination of conditioning medications (h-ATG, busulfan) and total body irradiation on the developing human fetus, including potential teratogenic or abortifacient effects.

If a study participant or partner of a male subject becomes pregnant or suspects she is pregnant, the participant should notify the study staff immediately. A female participant who becomes pregnant will be withdrawn from the study as outlined below. If a female participant or a partner of a male participant becomes pregnant, the participant will have contact follow-up with the study team to document the outcome of the pregnancy.

Because there is an unknown but potential risk for AEs in nursing infants secondary to the mother undergoing the study intervention, breastfeeding should be discontinued if the mother will undergo the study intervention.

Decisionally Impaired Adults: Adults who are unable to consent are eligible for enrollment in this protocol because they still benefit clinically from the study. However, the participant must have a DPA that can give consent. Similarly, enrolled participants who lose the ability to provide ongoing consent during study participation may continue in the study. The risks and benefits of participation for adults unable to consent should be identical to those described for less vulnerable patients.

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-26 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Engraftment rate of > 80% | six months and one year
  Engraftment rate of greater than or equal to 80% of patients achieving greater than or equal to 50% stable myeloid chimerism with or without the use of TBI.
Engraftment with no grade 3 GvHD | Day 100 and one year
  Engraftment as such should not occur with any Grade 3 or higher acute GvHD at Day 100 nor occurrence of extensive chronic GvHD

SECONDARY OUTCOMES:
Donor B cell engraftment | one year post transplant
  Attain donor B cell engraftment >50% donor chimerism with absolute number of B cells >80% of lower limit of normal
Donor T cell engraftment | one year post transplant
  Attain Donor T cell engraftment greater than or equal 30% donor chimerism with absolute number of T cells greater than or equal to 80% of lower limit of normal

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-I-0037.html